CLINICAL TRIAL: NCT02626403
Title: Effect of Fronto-parietal Transcranial Direct Stimulation on the Level of Consciousness in Patients With Disorders of Consciousness
Brief Title: Fronto-parietal tDCS in Severely Brain Injured Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, PhD, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/280
Record Dates: First submitted 2015-11-30; First posted 2015-12-10 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Vegetative State; Minimally Conscious State; Disorders of Consciousness
Keywords: vegetative state; minimally conscious state; disorder of consciousness; transcranial current direct stimulation; non invasive brain stimulation; neuromodulation
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS (Active Comparator): Patients will receive anodal tDCS (bilateral fronto-parietal stimulation) during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised) and neurophysiological assessment (8 channels EEG).
  Interventions: Device: Anodal tDCS
- sham tDCS (Sham Comparator): Patients will receive sham tDCS (15 second of stimulation) during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised) and neurophysiological assessment (8 channels EEG).
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — Patients will receive anodal tDCS during 20 minutes preceded and followed by a behavioral assessment (Coma Recovery Scale Revised) and an EEG. The anodes will be placed over F3, F4, CP5, and CP6 in order to stimulation the fronto-parietal cortex bilaterally.
  Arms: anodal tDCS
Device: Sham tDCS — Identical to anodal tDCS, except that the stimulation will be stopped after 15 seconds.
  Arms: sham tDCS

SUMMARY:
Previous studies showed that anodal transcranial direct current stimulation (tDCS) transiently improves performance of memory and attention. In severely brain injured patients with disorders of consciousness (DOC), a single stimulation over the left dorsolateral prefrontal cortex has shown to improve patients' sign of consciousness. Nevertheless, other brain areas could be stimulated in order to increase the number of responders. In this study, investigators will assess the effects of bilateral fronto-parietal tDCS on Coma Recovery Scale-Revised (CRS-R) scores in patients with DOC in a double-blind sham-controlled experimental design.

DETAILED DESCRIPTION:
Following severe brain damage and coma, some patients may remain in a vegetative state (VS) or minimally conscious state (MCS). At present, there are no evidence-based guidelines regarding the treatment of patients with disorders of consciousness (DOC). A previous study showed that a single stimulation (using transcranial direct current stimulation - tDCS) of the left prefrontal cortex induces an behavioral improvement in some patients in DOC. Nevertheless, only 43% of patients in MCS responded to the stimulation. Therefore, it is needed to find new protocols to increase the number of responders and improve the effect of tDCS in patients with DOC.

In this study, investigators aim to assess the effect of single session anodal (i.e., excitatory) transcranial direct current stimulation (tDCS) over right and left fronto-temporal cortices (using 4 anodes and 4 cathodes), on the level of consciousness of patients with DOC, in a double blind randomized sham controlled study. The anodes will be placed over F3, F3, CP5 and CP6.

tDCS is a form of safe non-invasive cortical stimulation, modulating cortical excitability under the electrodes, via weak polarizing currents. It has been reported that anodal tDCS transiently improves working memory and attention by stimulating the left DLPF in healthy subjects and patients with stroke, Parkinson's or Alzheimer's disease. By increasing the surface of the stimulated area, it is expected to increase the number of responders as patients' brain lesion are very heterogeneous and widespread.

ELIGIBILITY:
Inclusion Criteria:

* post comatose patients
* patients in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma
* patients < 28 days after the acute brain injury
* patients with a metallic cerebral implant
* cranioplasty
* shunt

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R total score | Baseline and directly after the tDCS (20 minutes)
  CRS-R will be performed before and after tDCS (anodal and sham). Comparison of the treatment effect (CRS-R total score after tDCS minus before) between real and sham tDCS

SECONDARY OUTCOMES:
Change in EEG | Baseline and directly after the tDCS (20 minutes)
  8 channels EEG will be record before and after tDCS to record potential cortical changes induce by the stimulation.
Change in CRS-R subscores | Baseline and directly after the tDCS (20 minutes)
  Same analysis as for CRS-R total score but on each of the 6 sub-scales

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Belgium

REFERENCES:
- [Result] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549